CLINICAL TRIAL: NCT01652313
Title: A Single Centre, Open-label, Multiple-dose Interventional Study Investigating the Pharmacokinetic Properties of Rasagiline (Lu 00-773) in Healthy Young Chinese Men and Women
Brief Title: Pharmacokinetic Properties of Rasagiline (Lu 00-773) in Healthy Young Chinese Men and Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13496A
Record Dates: First submitted 2012-07-23; First posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rasagiline (Experimental)
  Interventions: Drug: Rasagiline

INTERVENTIONS:
Drug: Rasagiline — 1 mg/day, tablets for 7 days, orally
  Other Names: Lu 00-773; Azilect®

SUMMARY:
The purpose of this study is to fulfil regulatory requirements for registration of a new chemical entity in China. Rasagiline is approved for the treatment of Parkinson's Disease (PD) in Europe and the US. Rasagiline is safe and well tolerated in healthy subjects, and the efficacy and safety has been demonstrated in placebo- and active comparator-controlled phase III studies.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a Chinese man or woman
* The subject is, in the opinion of the investigator, generally healthy
* If female, the subject must have a negative pregnancy test at screening and baseline, and agree not to try to become pregnant from Screening until after the Follow-up Visit

Exclusion Criteria:

* The subject is, in the opinion of the investigator, unlikely to comply with the clinical study protocol or is unsuitable for any other reason.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) AUC determination of rasagiline and its metabolite 1-aminoindan (1-AI) | 7 days
PK Cmax determination of rasagiline and its metabolite 1-aminoindan (1-AI) | 7 days

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- CN001, Beijing, China